CLINICAL TRIAL: NCT01031836
Title: A Phase II, Multicenter, Open-Label, Dose-Escalation Study to Evaluate Safety and Tolerability of IV or SC Dose of MEDI-545, a Fully Human Monoclonal Antibody Directed Against Interferon Alpha Subtypes, in Japanese Patients Who Have Systemic Lupus Erythematosus (SLE)
Brief Title: A Study to Evaluate Safety and Tolerability of IV or SC Dose of MEDI-545 in Patients With Systemic Lupus Erythematosus.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2800C00001
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Results first posted 2018-11-19 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Japanese; phase 2; safety; tolerability; MEDI-545; Autoimmune Disease; Immune System Diseases
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Immune System Diseases | interventions — sifalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- MEDI-545 1.0 mg/kg (Experimental): Cohort 1
  Interventions: Drug: MEDI-545
- MEDI-545 3.0 mg/kg (Experimental): Cohort 2
  Interventions: Drug: MEDI-545
- MEDI-545 10.0 mg/kg (Experimental): Cohort 3
  Interventions: Drug: MEDI-545
- MEDI-545 100 mg (Experimental): Cohort 4
  Interventions: Drug: MEDI-545
- MEDI-545 600 mg (Experimental): Cohort 5
  Interventions: Drug: MEDI-545 600
- MEDI-545 1,200 mg (Experimental): Cohort 6
  Interventions: Drug: MEDI-545

INTERVENTIONS:
Drug: MEDI-545 — Stage I: MEDI-545 1.0 mg/kg IV, on Day 1 and once every 2 weeks from Day 29, for a total of 14 doses.
  Stage II: MEDI-545 1.0 mg/kg IV once every 2 weeks for a total of 79 doses.
  Arms: MEDI-545 1.0 mg/kg
Drug: MEDI-545 — Stage I: MEDI-545 3.0 mg/kg IV, on Day 1 and once every 2 weeks from Day 29, for a total of 14 doses.
  Stage II: MEDI-545 3.0 mg/kg IV once every 2 weeks for a total of 79 doses
  Arms: MEDI-545 3.0 mg/kg
Drug: MEDI-545 — Stage I: MEDI-545 10.0 mg/kg IV, on Day 1 and once every 2 weeks from Day 29, for a total of 14 doses.
  Stage II: MEDI-545 10.0 mg/kg IV once every 2 weeks for a total of 79 doses.
  Arms: MEDI-545 10.0 mg/kg
Drug: MEDI-545 — Stage I: MEDI-545 100 mg SC, on Day 1 and weekly or once every 2 weeks from Day 29, for a total of 14 doses.
  Stage II: MEDI-545 100 mg SC once every 2 weeks for a total of 79 doses.
  Arms: MEDI-545 100 mg
Drug: MEDI-545 — Stage I: MEDI-545 1,200 mg IV once every 4 weeks from Day 1 for a total of 8 doses.
  Stage II: MEDI-545 1,200 mg IV once every 4 weeks for a total of 40 doses
  Arms: MEDI-545 1,200 mg
Drug: MEDI-545 600 — Stage I: MEDI-545 600 mg IV once every 4 weeks from Day 1 for a total of 8 doses.
  Stage II: MEDI-545 600 mg IV once every 4 weeks for a total of 40 doses.
  Arms: MEDI-545 600 mg

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability of MEDI-545 in Japanese adult SLE patients. This will be done by collecting the data from 3 cohorts of IV doses and 1 cohort of SC doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have previously met ≥4 of the 11 revised ACR criteria
* Have positive antinuclear antibody test (ANA) at ≥1:80 serum dilute in the past or at screening
* Have at least 1 system with a score of A or 2 systems with a score of B on the BILAG index at screening, or have a SELENA-SLEDAI score ≥6

Exclusion Criteria:

* Have received prednisone >20 mg/day (or an equivalent dose of another oral corticosteroid) within 14 days before Visit 2 (Day 1)
* Have received the following medications within 28 days before Visit 2 (Day 1):

  * Systemic cyclophosphamide at any dose
  * Cyclosporine at any dose
  * Tacrolimus at any dose
  * Thalidomide at any dose
  * Mycophenolate mofetil >2 g/day
  * Methotrexate >15 mg/week
  * Azathioprine >2 mg/kg/day
* Women who have a positive pregnancy test (serum hCG) at Visit 1

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-11-25 (Actual); Primary Completion 2012-11-07 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Takeuchi, Principal Investigator — Department of Internal Medicine School of Medicine Keio University; Yoshiya Tanaka, Principal Investigator — The University Hospital, University of Occupational and Environmental Health, Japan
Locations (7):
- Japan (7):
  - Research Site, Chiba
  - Research Site, Fukuoka
  - Research Site, Kanazawa
  - Research Site, Kawagoe-shi
  - Research Site, Kitakyushu-shi
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 7 centres in Japan. The first patient was enrolled on 25 November 2009 and the last enrolled patient had completed Stage II on 11 July 2016.
Pre-assignment Details: Thirty (30) patients received MEDI-545 either IV or SC treatment (5 patients in each cohort) at Stage I. Twenty-six (26) patients completed Stage I treatment and, out of these 26 patients, 21 patients were registered to continue in Stage II.
Groups:
- MEDI-545 1.0 mg/kg IV: MEDI-545 1.0 mg/kg IV once every 2 weeks
- MEDI-545 3.0 mg/kg IV: MEDI-545 3.0 mg/kg IV once every 2 weeks
- MEDI-545 10.0 mg/kg IV: MEDI-545 10.0 mg/kg IV once every 2 weeks
- MEDI-545 100 mg SC: MEDI-545 100 mg SC once every 2 weeks
- MEDI-545 600 mg IV: MEDI-545 600 mg IV once every 4 weeks
- MEDI-545 1200 mg IV: MEDI-545 1200 mg IV once every 4 weeks
Period: Stage I
Arm/Group | MEDI-545 1.0 mg/kg IV | MEDI-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100 mg SC | MEDI-545 600 mg IV | MEDI-545 1200 mg IV
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 3 | 5 | 5 | 5 | 4
Not Completed | 1 | 2 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 1
Period: Stage II
Arm/Group | MEDI-545 1.0 mg/kg IV | MEDI-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100 mg SC | MEDI-545 600 mg IV | MEDI-545 1200 mg IV
Started | 3 (1 patient who completed the study treatment in Stage I did not register in Stage II.) | 1 (2 patient who completed the study treatment in Stage I did not register in Stage II.) | 4 (1 patient who completed the study treatment in Stage I did not register in Stage II.) | 4 (1 patient who completed the study treatment in Stage I did not register in Stage II.) | 5 | 4
Completed | 1 | 1 | 2 | 1 | 3 | 3
Not Completed | 2 | 0 | 2 | 3 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 2 | 2 | 1 | 1
Not completed — Other | 2 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDI-545 1.0 mg/kg IV | MEDI-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100 mg SC | MEDI-545 600 mg IV | MEDI-545 1200 mg IV | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (3) | 43 (13) | 34 (9) | 37 (9) | 46 (10) | 48 (13) | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 5 | 5 | 4 | 28
  Male | 0 | 0 | 1 | 0 | 0 | 1 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Area Undre Curve (AUC) of MEDI-545 After First Dose in Stage I
Time Frame: After first dose in Stage I (0 upto 28 days)
Population: Pharmacokinetics (PK) populaton
Measure: Median (Full Range); unit: day*ug/mL
Groups:
- MEID-545 3.0 mg/kg IV: MEID-545 3.0 mg/kg IV once every 2 weeks
- MEDI-545 100mg SC: MEDI-545 100mg SC once every 2 weeks
- MEDI-545 600mg IV: MEDI-545 600mg IV once every 4 weeks
- MEDI-545 1200mg IV: MEDI-545 1200mg IV once every 4 weeks
Arm/Group | MEDI-545 1.0 mg/kg IV | MEID-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100mg SC | MEDI-545 600mg IV | MEDI-545 1200mg IV
Number analyzed (Participants) | 4 | 2 | 3 | 1 | 1 | 3
day*ug/mL | 261.98 (16.8) [226.18 to 332.80] | 647.93 (7.4) [614.06 to 681.80] | 3040.83 (24.2) [2284.94 to 3670.57] | 239.16 [239.16 to 239.16] | 2308.44 [2308.44 to 2308.44] | 5235.41 (11.6) [4646.86 to 5857.94]

2. Secondary Outcome: AUC0-14 of MEDI-545 After First Dose in Stage I
Description: Summary of area under the concentration-time curve from zero to Day 14.
Time Frame: After first dose in Stage I
Population: PK populaton
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | MEDI-545 1.0 mg/kg IV | MEID-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100mg SC | MEDI-545 600mg IV | MEDI-545 1200mg IV
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
day*ug/mL | 151.28 (19.3) | 432.26 (11.0) | 1728.01 (16.8) | 128.06 (56.1) | 1965.44 (41.4) | 4583.55 (15.2)

3. Primary Outcome: Number of Participants With Each Category of Adverse Events in Stage I
Time Frame: Stage I (up to 1 year)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-545 1.0 mg/kg IV | MEID-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100mg SC | MEDI-545 600mg IV | MEDI-545 1200mg IV
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Participants
  Any AE | 5 | 4 | 5 | 5 | 5 | 5
  Any AE of CTC grade at least 3 | 0 | 3 | 2 | 0 | 0 | 1
  Any AE with outcome=death | 0 | 0 | 0 | 0 | 0 | 0
  Any serious adverse events (SAE) | 0 | 3 | 3 | 0 | 0 | 3
  Any AE leading to discontinuation of IP | 1 | 1 | 1 | 0 | 0 | 0
  Any causally related AE | 5 | 3 | 5 | 3 | 4 | 5

4. Secondary Outcome: Maximum Observed Concentration (Cmax) of MEDI-545 After First Dose in Stage I
Time Frame: After first dose in Stage I
Population: PK populaton
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | MEDI-545 1.0 mg/kg IV | MEID-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100mg SC | MEDI-545 600mg IV | MEDI-545 1200mg IV
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
ug/mL | 29.04 (31.3) | 71.72 (19.6) | 311.17 (19.0) | 11.70 (61.1) | 244.54 (47.4) | 607.64 (16.1)

5. Secondary Outcome: Change From Baseline in 21-gene Signature Fold Change in Stage I
Description: 21-gene signature fold change is pharmacodynamics (PD) parameter measuring expression of type I IFN-inducible gene.
Time Frame: Stage I
Population: Safety population
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | MEDI-545 1.0 mg/kg IV | MEID-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100mg SC | MEDI-545 600mg IV | MEDI-545 1200mg IV
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
fold change
  Day 1 8 hours post-dose | -3.70 (2.07) | -5.68 (5.92) | -2.30 (0.93) | -1.17 (0.80) | -4.91 (2.26) | -3.44 (1.77)
  Day 3 | -2.57 (2.61) | -4.53 (7.02) | -2.49 (1.06) | -1.80 (0.97) | -4.81 (2.63) | -3.37 (1.69)
  Day 15 | -1.40 (2.56) | -1.11 (5.99) | -0.41 (1.60) | -0.59 (1.69) | -1.61 (1.23) | -1.84 (1.72)
  Day 29 | 0.03 (2.54) | -0.16 (8.44) | -0.34 (1.38) | -0.85 (0.81) | -1.13 (1.40) | -1.27 (2.46)

6. Secondary Outcome: Number of Participants With Positive Anti-drug Antibody (ADA) During Stage I
Time Frame: Stage I
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-545 1.0 mg/kg IV | MEID-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100mg SC | MEDI-545 600mg IV | MEDI-545 1200mg IV
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5
Participants | 0 | 1 | 0 | 0 | 0 | 1

7. Primary Outcome: Number of Participants in Each Category of Adverse Events (AE) in Stage II
Time Frame: Stage II (1 year to 3.5 years after first dose)
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | MEDI-545 1.0 mg/kg IV | MEID-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100mg SC | MEDI-545 600mg IV | MEDI-545 1200mg IV
Number analyzed (Participants) | 3 | 1 | 4 | 4 | 5 | 4
Participants
  Any AE | 3 | 1 | 4 | 4 | 5 | 4
  Any AE of CTC grade at least 3 | 0 | 0 | 1 | 2 | 3 | 2
  Any AE with outcome=death | 0 | 0 | 0 | 0 | 0 | 0
  Any serious adverse events (SAE) | 0 | 0 | 2 | 4 | 2 | 4
  Any AE leading to discontinuation of IP | 0 | 0 | 1 | 3 | 1 | 1
  Any causally related AE | 2 | 1 | 3 | 4 | 5 | 4

ADVERSE EVENTS:
Time Frame: Upto 1 year after treatment start for Stage I, 1 year to 3.5 years after treatment start for Stage II
Arm/Group | MEDI-545 1.0 mg/kg IV | MEDI-545 3.0 mg/kg IV | MEDI-545 10.0 mg/kg IV | MEDI-545 100 mg SC | MEDI-545 600 mg IV | MEDI-545 1200 mg IV
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/5 | 0/5 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 3/5 | 3/5 | 4/5 | 2/5 | 5/5
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5 | 5/5 | 5/5 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | MEDI-545 1.0 mg/kg IV (N=5) | MEDI-545 3.0 mg/kg IV (N=5) | MEDI-545 10.0 mg/kg IV (N=5) | MEDI-545 100 mg SC (N=5) | MEDI-545 600 mg IV (N=5) | MEDI-545 1200 mg IV (N=5)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Study Period: Stage I
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1 — Study Period: Stage I
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Study Period: Stage I
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 — Study Period: Stage I
Auditory disorders (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 — Study Period: Stage I
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 — Study Period: Stage I
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0/3 | 0/1 | 0/4 | 2/4 | 1 | 1/4 — Study Period: Stage II
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Bronchitis (Infections and infestations) | 0/3 | 0/1 | 0/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Pneumonia (Infections and infestations) | 0/3 | 0/1 | 0/4 | 0/4 | 1 | 0/4 — Study Period: Stage II
Pneumonia pneumococcal (Infections and infestations) | 0/3 | 0/1 | 0/4 | 0/4 | 1 | 0/4 — Study Period: Stage II
Pyelonephritis (Infections and infestations) | 0/3 | 0/1 | 0/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Sepsis (Infections and infestations) | 0/3 | 0/1 | 0/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Acute myocardial infarction (Cardiac disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 1 | 0/4 — Study Period: Stage II
Prinzmetal angina (Cardiac disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Cardiac ventricular thrombosis (Cardiac disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 1 | 0/4 — Study Period: Stage II
Cataract (Eye disorders) | 0/3 | 0/1 | 1/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Splenic infarction (Blood and lymphatic system disorders) | 0/3 | 0/1 | 0/4 | 1/4 | 0 | 0/4 — Study Period: Stage II
Dental caries (Gastrointestinal disorders) | 0/3 | 0/1 | 0/4 | 1/4 | 0 | 0/4 — Study Period: Stage II
Budd-Chiari syndrome (Hepatobiliary disorders) | 0/3 | 0/1 | 0/4 | 1/4 | 0 | 0/4 — Study Period: Stage II
Cerebral infaraction (Nervous system disorders) | 0/3 | 0/1 | 1/4 | 0/4 | 0 | 0/4 — Study Period: Stage II
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0/3 | 0/1 | 0/4 | 1/4 | 0 | 0/4 — Study Period: Stage II
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 1 | 0/4 — Study Period: Stage II
Hip arthroplasty (Surgical and medical procedures) | 0/3 | 0/1 | 0/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Deep vein thrombosis (Vascular disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 1 | 0/4 — Study Period: Stage II
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MEDI-545 1.0 mg/kg IV (N=5) | MEDI-545 3.0 mg/kg IV (N=5) | MEDI-545 10.0 mg/kg IV (N=5) | MEDI-545 100 mg SC (N=5) | MEDI-545 600 mg IV (N=5) | MEDI-545 1200 mg IV (N=5)
Nasopharyngitis (Infections and infestations) | 2 | 4 | 3 | 3 | 4 | 2 — Study Period: Stage I
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 1 — Study Period: Stage I
Otitis media (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 — Study Period: Stage I
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1 | 1 | 0 | 0 — Study Period: Stage I
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 0 — Study Period: Stage I
Dental caries (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 — Study Period: Stage I
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 — Study Period: Stage I
Headache (Nervous system disorders) | 0 | 1 | 3 | 0 | 1 | 0 — Study Period: Stage I
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 — Study Period: Stage I
Fatigue (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 — Study Period: Stage I
Pyrexia (General disorders) | 0/3 | 0/1 | 0/4 | 1/4 | 1 | 1/4 — Study Period: Stage II
Nasopharyngitis (Infections and infestations) | 3/3 | 1/1 | 2/4 | 3/4 | 4 | 3/4 — Study Period: Stage II
Upper respiratory tract infection (Infections and infestations) | 1/3 | 0/1 | 1/4 | 1/4 | 0 | 2/4 — Study Period: Stage II
Gastroenteritis (Infections and infestations) | 0/3 | 0/1 | 1/4 | 0/4 | 2 | 1/4 — Study Period: Stage II
Influenza (Infections and infestations) | 0/3 | 1/1 | 0/4 | 2/4 | 1 | 0/4 — Study Period: Stage II
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0/3 | 1/1 | 0/4 | 1/4 | 1 | 0/4 — Study Period: Stage II
Diarrhoea (Gastrointestinal disorders) | 1/3 | 0/1 | 0/4 | 1/4 | 1 | 0/4 — Study Period: Stage II
Gastritis (Gastrointestinal disorders) | 1/3 | 0/1 | 1/4 | 0/4 | 0 | 1/4 — Study Period: Stage II
Nausea (Gastrointestinal disorders) | 0/3 | 0/1 | 1/4 | 1/4 | 1 | 0/4 — Study Period: Stage II
Headache (Nervous system disorders) | 1/3 | 0/1 | 1/4 | 1/4 | 1 | 1/4 — Study Period: Stage II
Dizziness (Nervous system disorders) | 1/3 | 0/1 | 0/4 | 2/4 | 0 | 0/4 — Study Period: Stage II
Hypoaesthesia (Nervous system disorders) | 1/3 | 0/1 | 1/4 | 0/4 | 1 | 0/4 — Study Period: Stage II
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0/3 | 0/1 | 0/4 | 1/4 | 0 | 2/4 — Study Period: Stage II
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1/3 | 1/1 | 0/4 | 1/4 | 2 | 0/4 — Study Period: Stage II
Anaemia (Blood and lymphatic system disorders) | 0/3 | 0/1 | 0/4 | 0/4 | 2 | 1/4 — Study Period: Stage II

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No